CLINICAL TRIAL: NCT00420667
Title: Effect of Low Molecular Weight Heparin vs Unfractionated Heparin on Bleeding After Cardiac Surgery
Brief Title: Low Molecular Weight Heparin vs Unfractionated Heparin at Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Raffaele De Caterina, Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2007-01

CONDITIONS: Coronary Disease; Coronary Artery Bypass Grafting
Keywords: unfractionated heparin; enoxaparin; low molecular weight heparin; bypass surgery; bleeding
MeSH Terms: conditions — Coronary Disease; Hemorrhage | interventions — Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin

SUMMARY:
Because the impairment of platelet function may cause excess peri-operative bleeding, pre-operative aspirin discontinuation and heparin bridging are common at cardiac surgery. We aimed to evaluate the impact of a low-molecular-weight-heparin (LMWH), enoxaparin, and unfractionated heparin (UFH) on coagulation parameters and peri-operative bleeding in patients undergoing elective coronary artery bypass grafting (CABG) surgery after aspirin discontinuation.

The specific hypothesis of this study was that a 12 h interval is sufficient not to cause excess peri-operative bleeding, and is therefore an optimal compromise between antithrombotic efficacy and haemorrhagic safety.

DETAILED DESCRIPTION:
Since LMWH provide many pharmacokinetic advantages compared with UFH, and since they are a valid substitution for UFH in a number of settings, such as non-ST elevation acute coronary syndromes and prevention of venous thromboembolism, LMWH may provide a useful bridge to revascularization after aspirin discontinuation in patients undergoing CABG surgery. Obstacles to the spreading of this practice are mainly the absence of solid evidence of equivalence (or superiority) as to efficacy in this setting, and the proof of equal safety, namely the absence of excess bleeding because some studies have suggested an increased number of haemorrhagic complications after LMWH, particularly with the use of higher doses. This might here be a problem, as patients are here generally at high risk of thrombotic events and for this reason need higher doses than for prevention of venous thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 35-75 years with 3-vessel coronary artery disease (CAD)
* Candidates to elective CABG

Exclusion Criteria:

* Other additional (valve, carotid, etc.) simultaneous surgery required,
* Off-pump surgery,
* Any altered liver and kidney laboratory parameters,
* A history of any haemorrhagic disorders,
* Platelet count <100,000 and >450.000/μL,
* Treatment with ticlopidine or clopidogrel in the last month.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-11 (Actual); Primary Completion 2005-03 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Haemoglobin Concentration
Haematocrit
Platelet count
Transfusion Units

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Caterina, MD, PhD, Principal Investigator — Institute of Cardiology - G. d'Annunzio University, Chieti
Locations (1):
- Institute of Cardiology - S. Camillo Hospital, Chieti, CH, Italy

REFERENCES:
- [Background] Eagle KA, Guyton RA, Davidoff R, Edwards FH, Ewy GA, Gardner TJ, Hart JC, Herrmann HC, Hillis LD, Hutter AM Jr, Lytle BW, Marlow RA, Nugent WC, Orszulak TA; American College of Cardiology; American Heart Association. ACC/AHA 2004 guideline update for coronary artery bypass graft surgery: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1999 Guidelines for Coronary Artery Bypass Graft Surgery). Circulation. 2004 Oct 5;110(14):e340-437. No abstract available. PMID 15466654
- [Background] Goldman S, Zadina K, Moritz T, Ovitt T, Sethi G, Copeland JG, Thottapurathu L, Krasnicka B, Ellis N, Anderson RJ, Henderson W; VA Cooperative Study Group #207/297/364. Long-term patency of saphenous vein and left internal mammary artery grafts after coronary artery bypass surgery: results from a Department of Veterans Affairs Cooperative Study. J Am Coll Cardiol. 2004 Dec 7;44(11):2149-56. doi: 10.1016/j.jacc.2004.08.064. PMID 15582312
- [Background] Mangano DT; Multicenter Study of Perioperative Ischemia Research Group. Aspirin and mortality from coronary bypass surgery. N Engl J Med. 2002 Oct 24;347(17):1309-17. doi: 10.1056/NEJMoa020798. PMID 12397188
- [Background] Dacey LJ, Munoz JJ, Johnson ER, Leavitt BJ, Maloney CT, Morton JR, Olmstead EM, Birkmeyer JD, O'Connor GT; Northern New England Cardiovascular Disease Study Group. Effect of preoperative aspirin use on mortality in coronary artery bypass grafting patients. Ann Thorac Surg. 2000 Dec;70(6):1986-90. doi: 10.1016/s0003-4975(00)02133-0. PMID 11156107
- [Background] Ferraris VA, Ferraris SP. 1988: Preoperative aspirin ingestion increases operative blood loss after coronary artery bypass grafting. Updated in 1995. Ann Thorac Surg. 1995 Apr;59(4):1036-7. doi: 10.1016/0003-4975(95)00023-e. No abstract available. PMID 7695387
- [Background] Karthik S, Grayson AD, McCarron EE, Pullan DM, Desmond MJ. Reexploration for bleeding after coronary artery bypass surgery: risk factors, outcomes, and the effect of time delay. Ann Thorac Surg. 2004 Aug;78(2):527-34; discussion 534. doi: 10.1016/j.athoracsur.2004.02.088. PMID 15276512
- [Background] Sethi GK, Copeland JG, Goldman S, Moritz T, Zadina K, Henderson WG. Implications of preoperative administration of aspirin in patients undergoing coronary artery bypass grafting. Department of Veterans Affairs Cooperative Study on Antiplatelet Therapy. J Am Coll Cardiol. 1990 Jan;15(1):15-20. doi: 10.1016/0735-1097(90)90168-o. PMID 2404046
- [Background] Sirvinskas E, Veikutiene A, Grybauskas P, Cimbolaityte J, Mongirdiene A, Veikutis V, Raliene L. Influence of aspirin or heparin on platelet function and postoperative blood loss after coronary artery bypass surgery. Perfusion. 2006 Jan;21(1):61-6. doi: 10.1191/0267659106pf845oa. PMID 16485701
- [Background] Hirsh J, Raschke R. Heparin and low-molecular-weight heparin: the Seventh ACCP Conference on Antithrombotic and Thrombolytic Therapy. Chest. 2004 Sep;126(3 Suppl):188S-203S. doi: 10.1378/chest.126.3_suppl.188S. PMID 15383472
- [Background] Petersen JL, Mahaffey KW, Hasselblad V, Antman EM, Cohen M, Goodman SG, Langer A, Blazing MA, Le-Moigne-Amrani A, de Lemos JA, Nessel CC, Harrington RA, Ferguson JJ, Braunwald E, Califf RM. Efficacy and bleeding complications among patients randomized to enoxaparin or unfractionated heparin for antithrombin therapy in non-ST-Segment elevation acute coronary syndromes: a systematic overview. JAMA. 2004 Jul 7;292(1):89-96. doi: 10.1001/jama.292.1.89. PMID 15238596
- [Background] Clark SC, Vitale N, Zacharias J, Forty J. Effect of low molecular weight heparin (fragmin) on bleeding after cardiac surgery. Ann Thorac Surg. 2000 Mar;69(3):762-4; discussion 764-5. doi: 10.1016/s0003-4975(99)01366-1. PMID 10750757
- [Background] Prandoni P. Heparins and venous thromboembolism: current practice and future directions. Thromb Haemost. 2001 Jul;86(1):488-98. PMID 11487039
- [Background] Mismetti P, Laporte S, Darmon JY, Buchmuller A, Decousus H. Meta-analysis of low molecular weight heparin in the prevention of venous thromboembolism in general surgery. Br J Surg. 2001 Jul;88(7):913-30. doi: 10.1046/j.0007-1323.2001.01800.x. PMID 11442521
- [Background] Jones HU, Muhlestein JB, Jones KW, Bair TL, Lavasani F, Sohrevardi M, Horne BD, Doty D, Lappe DL. Preoperative use of enoxaparin compared with unfractionated heparin increases the incidence of re-exploration for postoperative bleeding after open-heart surgery in patients who present with an acute coronary syndrome: clinical investigation and reports. Circulation. 2002 Sep 24;106(12 Suppl 1):I19-22. PMID 12354703
- [Background] Burger W, Chemnitius JM, Kneissl GD, Rucker G. Low-dose aspirin for secondary cardiovascular prevention - cardiovascular risks after its perioperative withdrawal versus bleeding risks with its continuation - review and meta-analysis. J Intern Med. 2005 May;257(5):399-414. doi: 10.1111/j.1365-2796.2005.01477.x. PMID 15836656
- [Background] Sun JC, Crowther MA, Warkentin TE, Lamy A, Teoh KH. Should aspirin be discontinued before coronary artery bypass surgery? Circulation. 2005 Aug 16;112(7):e85-90. doi: 10.1161/CIRCULATIONAHA.105.546697. No abstract available. PMID 16103244